CLINICAL TRIAL: NCT04322136
Title: The Australasian Malignant PLeural Effusion (AMPLE) Trial - 3: A Randomised Study of the Relative Benefits of Combined Indwelling Pleural Catheter (IPC) and Talc Pleurodesis Therapy or Video-Assisted Thoracoscopic Surgery (VATS) in the Management of Patients With Malignant Pleural Effusion.
Brief Title: AMPLE-3: IPC Plus Talc vs VATS in Management of Malignant Pleural Effusion
Acronym: AMPLE-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Western Australia (Other)
Collaborators: Sir Charles Gairdner Hospital (Other); Fiona Stanley Hospital (Other); The Sutherland and St George Hospitals, Australia (Unknown); Hollywood Private Hospital, Australia (Unknown); Wellington Hospital (Other Government); Northern Hospital, Australia (Other); Concord Hospital (Other); Royal Adelaide Hospital, Australia (Unknown); St John of God Midland Hospital, Australia (Unknown); St John of God Murdoch Hospital, Australia (Unknown); Westmead Hospital, Australia (Unknown); St Vincent's Hospital Melbourne (Other); The Prince Charles Hospital (Other Government); Sunshine Coast Hospital and Health Service (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Toronto General Hospital (Other); Universiti Kebangsaan Malaysia Medical Centre (Other); Hospital Queen Elizabeth, Malaysia (Other Government); Johns Hopkins University (Other); John Hunter Hospital (Other Government); Wesley Hospital, Australia (Unknown); Auckland City Hospital (Other Government); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, YC Gary Lee, Professor, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMPLE-3; ACTRN12618001013257 (Other: ANZCTR)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Malignant Pleural Effusion; Respiratory Disease; Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Respiration Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPC (with talc pleurodesis if suitable) (Other): The patients will undertake daily drainage to day 14 post insertion. The drainage will either be performed by the participant's carer or nurses in the community. A bottle or bag will be attached to the drain to allow for removal of accumulated pleural fluid. Once completed the drain will be reattached to the pleural catheter.
  Participants will be taught how to perform pleural drainage by the main study doctor at the hospital or a specialist nurse. They will drain their own IPCs at home with the either the help of a family member or friend or have access to community nursing support systems.
  Interventions: Device: Indwelling pleural catheter (with talc pleurodesis if suitable)
- Pleurodesis via VATS (Other): Participants will undergo VATS within two weeks of randomisation. VATS is usually performed in an operating theatre, using either general anaesthesia or local anaesthesia with sedation. The pleural fluid will be removed and adhesions can be divided (adhesiolysis). Assessment of lung re-expansion will be performed intra-operatively. If lung re-expansion is adequate (as judged by the operating surgeon), a variety of techniques may be employed to induce a pleurodesis, including, but not limited to, talc poudrage and mechanical abrasion. Decortication may be performed if deemed appropriate and feasible by the operating surgeon. A chest drain will be left in situ after the surgery. Post-operative care will be administered as per local practice.
  Interventions: Procedure: Pleurodesis via Video-assisted thoracoscopic surgery

INTERVENTIONS:
Procedure: Pleurodesis via Video-assisted thoracoscopic surgery — Video-assisted thoracoscopic surgery is a type of key-hole surgery performed under general anaesthetic and usually single lung ventilation by a cardio-thoracic surgeon. This is expected to take about 1 hour. Between one and three ports are used to insert a camera and instruments into the chest cavity. Adhesions can be broken down if present and the lining of the lung (visceral pleura) can sometimes be removed (decortication) to facilitate lung re-expansion. The surgeon can then perform either mechanical abrasion or talc poudrage to induce inflammation and subsequent pleurodesis. A chest drain is left in situ post-operatively and is removed when the fluid draining is below a certain volume depending on local practice.
  Arms: Pleurodesis via VATS
Device: Indwelling pleural catheter (with talc pleurodesis if suitable) — Once the indwelling pleural catheter is inserted, the pleural fluid will be evacuated as completely as possible. If the lung fully re-expands, 4-5g of sterile graded talc will be instilled via the IPC. The participant will then be discharged on a daily drainage regimen for 14 days. At review in clinic on day 14, the participant will be assessed for spontaneous pleurodesis (<50ml drainage on 3 consecutive drainage attempts). If pleurodesis has occurred and there is no residual symptomatic effusion, arrangements will be made for IPC removal. Otherwise the participant will switch to a symptom-guided drainage regimen. If the lung does not fully re-expand following complete fluid evacuation, they will be discharged on a symptom-guided regimen without instillation of talc. The drainage regimen will continue for the duration of the study and beyond if pleurodesis has not occurred and pleural fluid continues to accumulate.
  Arms: IPC (with talc pleurodesis if suitable)

SUMMARY:
The purpose of this study is to determine if an indwelling catheter is more effective than surgical pleurodosis in treating malignant pleural effusion.

Who is it for?

You may be eligible for this study if you are an adult who is suffering from symptomatic proven pleural malignancy or an otherwise unexplained pleural effusion.

Study details

Consenting participants will be randomised to one of two treatment arms:

* Arm 1: Indwelling pleural catheter. A long term catheter is inserted under the skin in order to allow ongoing drainage of the pleural fluid. Participants will then be instructed to undergo a daily drainage regimen for 14 days at home.
* Arm 2: Surgical pleurodesis. Participants under a key-hole surgery to remove fluid and facilitate lung re-expansion.

Participants will then be followed up at discharge, 14 days, monthly for 6 months and then every 3 months up to one year post-procedure. These visits will include completion of Quality of Life questionnaires, a chest xray, an ultrasound (if thought necessary) and if you are at the lead site (Sir Charles Gairdner Hospital) a review of your Actigraphy logs up to 6 months after discharge.

It is hoped this research will help to provide effective symptom control with minimal intervention for those with malignant pleural effusion.

DETAILED DESCRIPTION:
Participants will be randomly assigned (1:1) to one of two arms:

Arm 1: Indwelling pleural catheter (with talc pleurodesis if suitable) Arm 2: Pleurodesis via Video-assisted thoracoscopic surgery

Arm 1: Indwelling pleural catheter is a long-term catheter that is tunnelled under the skin and allows ongoing drainage of pleural fluid by the patient or carer at home. It is inserted using local anaesthetic with or without sedation depending on local practice. An experienced respiratory physician inserts the catheter. Once the catheter is inserted, the pleural fluid will be evacuated as completely as possible. If the lung fully re-expands and there is no contraindication to talc pleurodesis, 4-5g of sterile graded talc will be instilled via the IPC. The participant will then be discharged on a daily drainage regimen for 14 days. The drainage will either be performed by the participant's carer or nurses in the community. A bottle or bag will be attached to the drain to allow for removal of accumulated pleural fluid. Once completed the drain will be reattached to the pleural catheter. At review in clinic on day 14 (+/- 2 days), the participant will be assessed for spontaneous pleurodesis (<50ml drainage on 3 consecutive drainage attempts). If pleurodesis has occurred and there is no residual symptomatic effusion, arrangements will be made for IPC removal. Otherwise the participant will switch to a symptom-guided drainage regimen. If the lung does not fully re-expand following complete fluid evacuation, they will be discharged on a symptom-guided regimen without instillation of talc. The drainage regimen will continue for the duration of the study and beyond if pleurodesis has not occurred and pleural fluid continues to accumulate. All participants will remain under the care of their study doctors who are also their usual physicians, after the end of the study.

Arm 2: Video-assisted thoracoscopic surgery is a type of key-hole surgery performed under general anaesthetic and usually single lung ventilation by a cardio-thoracic surgeon. This is expected to take about 1 hour. Between one and three ports are used to insert a camera and instruments into the chest cavity. Adhesions can be broken down if present and the lining of the lung (visceral pleura) can sometimes be removed (decortication) to facilitate lung re-expansion. The surgeon can then perform either mechanical abrasion or talc poudrage to induce inflammation and subsequent pleurodesis. A chest drain is left in situ post-operatively and is removed when the fluid draining is below a certain volume depending on local practice.

Participants in both arms will be reviewed at the same time points - at discharge, 14 days post-procedure, monthly to 6 months, then 3-monthly to 1 year. The reviews will include quality of life and breathlessness questionnaires.

All data will be obtained by the designated study research team who will carry out the IPC insertions and where VATs pleurodesis is undertaken, the research team will liaise directly with the study surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a symptomatic MPE*
2. Predicted survival of more than 6 months
3. Eastern Cooperative Oncology Group (ECOG) score = Peformance status defined as a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc. ECOG 0-1 (or ECOG greater than or equal to 2 if it is felt that removal of pleural fluid would improve their status to 0 or 1).

   * MPE is defined as histologically/cytologically proven pleural malignancy or an otherwise unexplained pleural effusion in the context of clinically proven cancer elsewhere.

Exclusion Criteria:

1. Age <18yrs;
2. Unfit to undergo a surgical procedure (American Society of Anaesthesiologists Score >/=4); 3. Pleural infection;

4. Chylothorax; 5. Pregnancy or lactation; 6. Uncorrectable bleeding diathesis; 7. Previous ipsilateral lobectomy/pneumonectomy; 8. Inability to consent or comply with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Need for an ipsilateral pleural intervention | Participants will be followed for a maximum of 12 months or until death if sooner.
  Proportion of participants requiring an ipsilateral (on the same side) pleural procedure for management of symptomatic re-accumulation of pleural fluid including surgical procedure, chest drain insertion, attempted therapeutic thoracentesis. This is a composite outcome.
  Data will be obtained from the participants and the hospital record.

SECONDARY OUTCOMES:
Need for repeat ipsilateral pleural intervention including diagnostic aspiration | The study is for 12 months or until death if prior.
  Proportion of participants requiring an ipsilateral pleural procedure including diagnostic aspirate.
  Data will be obtained from the participants and the hospital record.
Time to symptomatic effusion recurrence | The study is for 12 months or until death if prior.
  Time to effusion recurrence - will be assessed using chest x-ray and ultrasound at each visit. Recurrent effusion is defined as greater than 25% opacity on chest x-ray on the side of the intervention as judged by two independent clinicians and evidence of pleural fluid on ultrasound.
All-cause hospital days | The study is for 12 months or until death if prior.
  Length of stay post-procedure and hospitalization for any cause (except for elective admissions for chemotherapy) will be recorded for all patients post randomisation. Admissions will be analysed as total admission days and also pleural-related admission days.
  The data will be collected from participants and the hospital records.
Degree of breathlessness | Scores will be recorded daily for 28 days, then monthly to 6 months and 3-monthly until 12 months.
  Degree of breathlessness will be measured by a 100mm Visual Analogue Scale (VAS). The VAS is a 100mm line anchored with "no breathlessness" at 0mm and "worst breathlessness imaginable" at 100mm.
Pain scale | Scores will be recorded daily for 28 days, monthly to 6 months and then 3-monthly to 12 months
  Pain will be assessed using a 100mm visual analogue scale. The 100mm horizontal line will be anchored with "no pain" at 0mm and "worst pain imaginable" at 100mm.
Quality of Life (QoL) | QoL will be measured at baseline, day 7-10 post-procedure, then monthly to 6 months then 3 monthly to 12 months.
  Quality of Life (QoL) will be measured using two instruments: EQ-5D-5L is a standardised measure of HRQoL that comprises five dimensions including mobility, self-care, usual activities, pain//discomfort and anxiety/depression. VAS QoL records self-rated health on a 100mm line anchored with "best imaginable health state" at 0mm and "worst imaginable health state" at 100mm.
Physical activity patterns | Monthly to 12 months at lead site only.
  Actigraphy is one part of the study and is an outcome comprising a few different factors. Physical activity patterns, vigorous activity and periods of sedentary behaviour, will be evaluated by a well validated triaxial accelerometer (ActiGraph GT3X+, Pensacola, FL, USA). Objective physical activity patterns will be assessed by 7-day triaxial accelerometer assessment providing an indication of functional status. The Actigraph device is reliable, with excellent test-retest reproducibility in cancer research and rated as 'user friendly' by both healthy and patient populations.
Adverse events from time of enrolment | Assessed continuously up to 12 months.
  Adverse events from randomization until end of follow-up or death. An adverse event is defined as any participant-reported or medical records complications associated with the IPC or VATS pleurodesis, such as pleural infection, cellulitis, pain, symptomatic loculation, tube blockage, catheter tract metastases, parenchymal air leak etc., and any peri/post-procedural complications such as prolonged air-leak, atelectasis, pneumonia, cardiovascular complications, acute kidney injury or drop in haemoglobin requiring transfusion.
Overall survival from randomisation. | From randomisation up to 12 months
  Overall Survival will be recorded from date of enrolment to death or end of study follow-up. Survival difference between IPC and VATS management of malignant pleural effusion has not been previously studied.
Pleural-related hospital days. | The study is for 12 months or until death if prior.
  Pleural-related hospital days. Length of stay post-procedure and hospitalization for any cause (except for elective admissions for chemotherapy) will be recorded for all patients post randomisation. Admissions will be analysed as total admission days and also pleural-related admission days.
  The data will be collected from participants and the hospital records.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Respiratory Health, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No